CLINICAL TRIAL: NCT00720616
Title: Effects of a Fixed Low Dose Growth Hormone Therapy on Insulin Sensitivity, Metabolic Profile, Adipocyte IGF-I and Insulin Signalling, Intramyocellular and Intrahepatic Lipids, and Cortisol Metabolism in Subjects With Metabolic Syndrome.
Brief Title: Low Dose Growth Hormone Treatment in Subjects With Metabolic Syndrome.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kevin Yuen, Associate Professor of Endocrinology, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB4481
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Metabolic Syndrome
Keywords: Growth hormone; Metabolic syndrome; Insulin sensitivity
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — Human Growth Hormone; Growth Hormone; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Growth hormone or Placebo 0.1 mg/day self-administrated once a day.
  Interventions: Drug: Norditropin

INTERVENTIONS:
Drug: Norditropin — Norditropin 0.1 mg/day self-administered once a day subcutaneously
  Other Names: Growth hormone, metabolic syndrome, insulin sensitivity

SUMMARY:
Study hypothesis:

Low dose growth hormone (GH), through its generation of free 'bioavailable' insulin-like growth factor (IGF)-I, can improve insulin sensitivity and the metabolic profile of subjects with metabolic syndrome.

Study aims:

The purpose of this study is to determine the mechanism of how low dose GH treatment affects the body's sensitivity to insulin actions and whether this low GH dose can affect the body's handling of steroid hormone levels (cortisol clearance) and fat deposition in subjects with metabolic syndrome.

Study design: Subjects that satisfy the criteria of metabolic syndrome (central obesity, treated or untreated high blood pressure, high cholesterol and impaired fasting glucose levels) will be invited to participate in this study. The subjects will be assessed at the initial visit to ascertain their suitability before further participation in the study. If eligible, an equal number of men and women will be randomized (like a flip of a coin) to receive either daily low dose GH or placebo injections first for 12 weeks, before exchanging over for another 12 weeks of treatment after a 4-week washout period. Before, during and after treatment, the subjects will be assessed at frequently with blood tests, scans and fat biopsies. During the study, the subjects will be studied 4 times at the Oregon Clinical and Translational Research Institute (OCTRI). At the first, second and final visit, testing will include scans to measure the amount of whole body fat and fat in the stomach area, muscle, and liver; blood tests to measure levels of cortisol, and fat tissue (taken from a biopsy) analysis to measure the density of insulin-like growth factor-I (a hormone stimulated by growth hormone in the body) in fat; whereas blood tests to examine how well insulin works in the body (insulin sensitivity) will be collected at all visits of the study.

DETAILED DESCRIPTION:
The study will be a double-blinded randomized placebo-controlled cross-over study. Thirty subjects will be screened for eligibility initially, and the first 12 eligible subjects will be enrolled. Six subjects will be randomized to receive the low GH dose (0.1 mg/day) treatment and 6 subjects to receive Placebo treatment for 12 weeks, exchanging their treatment for a further 12 weeks after a 4-week washout period. The study drugs will be stored at the Oregon Health and Science University (OHSU) Research Pharmacy and following randomization, the subjects will be taught by either the Principal Investigator or one of our Endocrine Nurses to self-administer the injections using Norditropin/Placebo vials and insulin syringes into the abdomen at 2200h. Randomization for treatment assignment will be performed by an investigator not directly involved in the patients' recruitment, treatment and follow-up care. The randomization process will be performed by computerized pre-assigned random codes by blocks, stratified by age and examined for possible differences in body mass index. During their in-patient stay at the Oregon Clinical and Translational Research Institute (OCTRI) at OHSU, subjects will only be allowed to eat the food provided to them by the OCTRI.

Initial Screening Assessment (outpatient)

The following assessments will be performed:

* Written informed consent
* Demographics (demographic information including the subject's birth date, and race)
* Physical exam and medical history
* Previous/significant medical history
* Concomitant medication review
* Vital signs, e.g., pulse and blood pressure measurements
* Height, weight and waist circumference
* Laboratory findings, e.g. CBC, electrolytes, and fasting glucose levels

Visit 1, Baseline Assessment for the First Treatment Phase (in-patient)

The following is a description of the assessments that will be performed after consent is obtained:

* Physical exam and medical history
* Vital signs, e.g., pulse and blood pressure measurements
* Height and weight
* Waist circumference measurement
* Concomitant medication review
* Urine pregnancy test for female child-bearing subjects
* Fasting blood assessments, e.g., hemoglobin, glucose, insulin, C-peptide, serum total and free IGF-I, IGFBP-3, C-reactive protein, non-esterified fatty acids (NEFAs), adiponectin, and ghrelin
* A 3-hour one-step hyperinsulinemic euglycemic clamp
* MRS and DEXA scans
* Cortisol clearance rate assessments
* Fat biopsy
* Randomization to GH or Placebo
* Teach GH or Placebo self-administration

Visit 2, Final Assessment for the First Treatment Phase (Week 12 +/- 1 week) (outpatient)

The following is a description of the assessments that will be performed at the end of the first treatment phase with either GH or Placebo. Subjects will also be monitored for safety with the collection of the following:

* Physical exam and medical history
* Vital signs, e.g. pulse and blood pressure measurements
* Height and weight
* Waist circumference measurement
* Concomitant medication review
* Adverse event recording
* Urine pregnancy test for female child-bearing subjects
* Fasting blood assessments, e.g., hemoglobin, glucose, insulin, C-peptide, serum total and free IGF-I, IGFBP-3, C-reactive protein, non-esterified fatty acids (NEFAs), adiponectin, and ghrelin
* A 3-hour one-step hyperinsulinemic euglycemic clamp
* MRS and DEXA scans
* Cortisol clearance rate assessments
* Fat biopsy

Washout Period and Crossover after the first treatment phase with GH or Placebo, the subjects will have a 4-week washout period and the treatment will be crossed over for another 12-week treatment phase with either GH or Placebo. During this time, the subjects will be advised to maintain a stable diet and weight.

Visit 3, Baseline Assessment for the Second Treatment Phase (Week 16 +/- 1 week) (as outpatient)

The following is a description of the assessments that will be performed:

* Physical exam and medical history
* Vital signs, e.g., pulse and blood pressure measurements
* Height and weight
* Waist circumference measurement
* Concomitant medication review
* Urine pregnancy test for female child-bearing subjects
* Fasting blood assessments, e.g., hemoglobin, glucose, insulin, C-peptide, serum total and free IGF-I, IGFBP-3, C-reactive protein, non-esterified fatty acids (NEFAs), adiponectin, and ghrelin
* A 3-hour one-step hyperinsulinemic euglycemic clamp
* MRS and DEXA scans
* Cortisol clearance rate assessments
* Fat biopsy
* Treatment exchanged to Placebo or GH

Visit 4, Final Assessment for the Second Treatment Phase (Week 28 +/- 1 week) (as inpatient)

The following is a description of the assessments that will be performed at the end of the second treatment phase with either GH or Placebo. Subjects will also be monitored for safety with the collection of the following:

* Physical exam and medical history
* Vital signs, e.g., pulse and blood pressure measurements
* Height and weight
* Waist circumference measurement
* Concomitant medication review
* Urine pregnancy test for female child-bearing subjects
* Fasting blood assessments, e.g., hemoglobin, glucose, insulin, C-peptide, serum total and free IGF-I, IGFBP-3, C-reactive protein, non-esterified fatty acids (NEFAs), adiponectin, and ghrelin
* A 3-hour one-step hyperinsulinemic euglycemic clamp
* MRS and DEXA scans
* Cortisol clearance rate assessments
* Fat biopsy

Because of the potentially long duration of Visits 1, 2 and 4, the studies can either be divided into two separate admissions upon prior arrangement or can be done all at once with one admission, depending on the subject's wishes and schedule.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Age 21 to 65 years
* Body mass index between 25 to 40 kg/m2
* Diagnosis of MBS based on the consensus statement by the International Diabetes Federation i.e., central obesity defined by waist circumference in men of ≥ 94 cm and in women of ≥ 80 cm plus two other components from the following: 1) dyslipidemia (triglyceride levels ≥ 150 mg/dl or on therapy and/or HDL in men of < 40 mg/dl and in women of < 50 mg/dl or on therapy); 2) hypertension (blood pressure ≥ 130/85 mmHg or on therapy and 3) hyperglycemia (fasting plasma glucose ≥ 100 mg/dl or on therapy)
* Stable weight and diet for at least 6 months prior to study entry
* Normal thyroid function
* Normal renal and hepatic function
* Able to self administer GH/Placebo injections

Exclusion Criteria:

* Inability to comply with study requirements
* Body mass index < 30 kg/m2 and > 40 kg/m2 (patients with body mass index > 40 kg/m2 are excluded because they will not fit into the MRS scanner)
* Untreated hypothyroidism or hyperthyroidism
* Anemia from any cause
* Known diabetes mellitus
* Patients with an increased risk of venous thrombosis or previous history of recurrent venous thrombosis
* Patient on any insulin-sensitizers (e.g., Metformin, Rosiglitazone, Pioglitazone) within 30 days of screening assessment
* Patient on any anti-androgens (e.g., Spironolactone, Cyproterone acetate, Flutamide, Finasteride) within 30 days of screening assessment
* Patient with other concurrent illnesses
* Pregnant (positive pregnancy test) prior enrollment in the study or planning to conceive whilst participating in the study
* Emotional/social instability likely to prejudice study completion
* Previous history of known malignancy
* Recurrent or severe unexplained hypoglycemia
* Known or suspected drug/alcohol abuse
* Patient with any metals in the body
* Any other condition/s that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Changes in insulin sensitivity, and adipocyte IGF-I and insulin receptor signaling. | 24 months

SECONDARY OUTCOMES:
Changes in body composition, cortisol production rates, and muscle and liver intramyocellular content. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C. Yuen, MRCP(UK), MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Yuen K, Wareham N, Frystyk J, Hennings S, Mitchell J, Fryklund L, Dunger D. Short-term low-dose growth hormone administration in subjects with impaired glucose tolerance and the metabolic syndrome: effects on beta-cell function and post-load glucose tolerance. Eur J Endocrinol. 2004 Jul;151(1):39-45. doi: 10.1530/eje.0.1510039. PMID 15248820
- See also: American Endocrine Society — http://www.endo-society.org/